CLINICAL TRIAL: NCT01674309
Title: Phase II: First Line Treatment by FOLFIRINOX for Patients With a Rectum Cancer With Synchronous Non Resectable Metastasis
Brief Title: First Line Treatment by FOLFIRINOX for Patients With a Rectum Cancer With Synchronous Non Resectable Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1102
Record Dates: First submitted 2012-04-02; First posted 2012-08-28 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2018-02

CONDITIONS: Adenocarcinoma of Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm study/ non randomized trial (Other): FOLFORINOX
  Interventions: Drug: FOLFORINOX

INTERVENTIONS:
Drug: FOLFORINOX — INTRAVENOUS administration

SUMMARY:
The FOLFIRINOX protocol seems a promising protocol as attack treatment of a rectum cancer, with an objective response rate of about 70 %. This phase II is to investigate if this systematic attack chemotherapy could control at the same time the rectal tumor and the synchronous metastasis without compromising secondarily the tumor or the metastasis resection or a radiochemotherapy administration.

1. The main objective of the trial is to investigate the tumoral control rate at 4 months, according to the RECIST criteria (version 1.1).
2. The secondary objectives are:

   * safety of the treament,
   * rate of local failure and local complication (occlusion, important bleedings, resistant pains with morphinic treatment, perforation),
   * survival without local failure (radiological or clinical progression of the rectal cancer or local complication),
   * rectal tumor response rate (CT scan, MRI and endocopy),
   * metastasis response rate,
   * disease free survival after complete resection (of primitive tumor and metastases),
   * progression free survival (local or distal),
   * overall survival, quality of life (QLQ-C30 + CR 29).

DETAILED DESCRIPTION:
The FOLFIRINOX protocol seems a promising protocol as attack treatment of a rectum cancer, with an objective response rate of about 70 %. This phase II is to investigate if this systematic attack chemotherapy could control at the same time the rectal tumor and the synchronous metastasis without compromising secondarily the tumor or the metastasis resection or a radiochemotherapy administration.

1. The main objective of the trial is to investigate the tumoral control rate at 4 months, according to the RECIST criteria (version 1.1).
2. The secondary objectives are:

   * safety of the treament,
   * rate of local failure and local complication (occlusion, important bleedings, resistant pains with morphinic treatment, perforation),
   * survival without local failure (radiological or clinical progression of the rectal cancer or local complication),
   * rectal tumor response rate (CT scan, MRI and endocopy),
   * metastasis response rate,
   * disease free survival after complete resection (of primitive tumor and metastases),
   * progression free survival (local or distal),
   * overall survival, quality of life (QLQ-C30 + CR 29).
3. Inclusion and non inclusion criteria
4. Treatment
5. Follow up

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the rectum, the lower pole less than 15 cm from the anal verge
* Patient should not have receive any treatment for cancer
* Synchronous metastases with unresectable hepatic and/or lung localization or uncertain resectability (potentially resectable)
* Measurable lesions by RECIST 1.1 (metastasis and primary cancer of the rectum)
* Age ≥ 18 years
* WHO ≤ 2
* ANC ≥ 1.5 x 10 9/L, platelets ≥ 100 x 10 9/L, creatinine clearance ≥ 60 mL/min
* Hemoglobin ≥ 10 g /dL
* Signed informed consent

Exclusion Criteria:

* Rectal Cancer in occlusion requiring surgery or a prosthesis in emergency
* Rectal bleeding severe and active
* Prior pelvic irradiation
* History of cancer, except non-melanoma skin cancer, carcinoma in situ of the cervix treated curatively and other cancers treated curatively if they do not relapse over 3 years,
* Hepatic impairment (total bilirubin> 1.5 x upper limit of normal (ULN) and serum albumin <25g / L); known Gilbert's disease
* Uncontrolled severe infection,
* Severe pain (VAS> 5/10) uncontrollable by opioid therapy
* Symptomatic sensorimotor peripheral neuropathy
* Pregnant or lactating patients or patient of both sexes with childbearing potential and not using adequate contraception method
* Patient receiving or having received an experimental therapy within 4 weeks prior to enter into the study or participating in another clinical study of other experimental drugs
* Known hypersensitivity to any component of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Tumor control rate of the primary tumor and metastasis | 4 months
  The tumor control rate of the primary site and metastasis is defined as Complete response or Partial response or stability according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Toxicity of the treatment | Up to 4 months after Last Patient First Visit
  Number of patients presenting the main toxicities during the study
rate of local failure and local complication (occlusion, important bleedings, resistant pains with morphinic treatment, perforation) | 4 months
  The rate is defined as the clinical progression or a radiological progression of the rectum cancer or a local complication due to the treatment or due to the progression
survival without local failure (radiological or clinical progression of the rectal cancer or local complication) | Up to 4 months after Last Patient First Visit
  The survival time is defined as the time between the patient's inclusion and the time of the local failure or patient's death
rectal tumor response rate (CT scan, MRI and endocopy) | 4 months
  The rectal tumor response rate is the Complete response or the Partial response of the rectal tumor using RECIST 1.1 criteria
metastasis response rate | 4 months
  The metastasis tumor response rate is the Complete response or the Partial response of metastasis using RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste BACHET, Dr, Principal Investigator — CHU de La Pitié Salpetrière - APHP
Locations (37):
- France (37):
  - CHU, Amiens
  - CHU, Angers
  - CH, Avignon
  - CH, Beauvais
  - CHU, Besançon
  - CH, Béziers
  - Avicennes, Bobigny
  - CHU - Ht Lévêque, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHU d'Estaing, Clermont-Ferrand
  - Colmar Ch, Colmar
  - Centre G.F. Leclerc, Dijon
  - CHU, Dijon
  - Polyclinique, Francheville
  - CHD Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHRU - Hôpital Huriez, Lille
  - CHU La Timone, Marseille
  - Ipc - Cac, Marseille
  - CH Layne, Mont-de-Marsan
  - Centre Cahterine de Sienne, Nantes
  - Polyclinique le Languedoc, Narbonne
  - CH Georges Menon, Niort
  - CHR - Gasto, Orléans
  - AP - HP - Pitié Salpêtrière, Paris
  - CH, Pau
  - CH, Perpignan
  - CHU, Rouen
  - CH Le Foll, Saint-Brieuc
  - Clinique Armoricaine, Saint-Brieuc
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - CH Robert Morlevat, Semur-en-Auxois
  - CAC, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - Hôpitaux du Leman, Thonon-les-Bains
  - Clinique Saint Jean du Languedoc, Toulouse
  - CHRU Trousseau, Tours

REFERENCES:
- [Result] Bachet JB, Lucidarme O, Levache CB, Barbier E, Raoul JL, Lecomte T, Desauw C, Brocard F, Pernot S, Breysacher G, Lagasse JP, Di Fiore F, Etienne PL, Dupuis OJM, Aleba A, Lepage C, Taieb J; for FFCD 1102 investigators. FOLFIRINOX as induction treatment in rectal cancer patients with synchronous metastases: Results of the FFCD 1102 phase II trial. Eur J Cancer. 2018 Nov;104:108-116. doi: 10.1016/j.ejca.2018.09.006. Epub 2018 Oct 18. PMID 30343254